CLINICAL TRIAL: NCT00403156
Title: A Phase I Study of the Inhibition of Platelet Derived Growth Factor Using Imatinib Mesylate Combined With Intravitreal Ranibizumab in the Treatment of Choroidal Neovascularization Secondary to Age-Related Macular Degeneration
Brief Title: Imatinib Mesylate Combined With Intravitreal Ranibizumab in the Treatment of Choroidal Neovascularization Secondary to Age-Related Macular Degeneration
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Richard Spaide, MD, Vitreous Retina Macula Consultants of New York
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF3989S
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Choroidal Neovascularization
Keywords: Macular Degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Imatinib Mesylate; Ranibizumab

INTERVENTIONS:
Drug: Imatinib Mesylate /Ranibizumab

SUMMARY:
The purpose of study is to determine if Lucentis combined with imatinib mesylate will help treatment in patients with newly diagnosed choroidal neovascularization.

DETAILED DESCRIPTION:
This is an open-label dose escalating study (n=15) to evaluate the safety and tolerability of the addition of imatinib mesylate to the Lucentis treatment regime over a 6 month period in patients with newly diagnosed choroidal neovascularization:

* 5 patients will be treated with 4 weeks of imatinib mesylate 400mg per day (the lowest typical starting dose) to be started concurrently with ranibizumab (Lucentis) 0.5mg intravitreal injection. The patients would be injected at monthly intervals for the first 3 months followed by treatment on an as needed basis.
* If imatinib mesylate is safely tolerated for the first 4 weeks, the following set of 5 patients will be treated with 6 weeks of imatinib mesylate 400mg per day to be started concurrently with Lucentis 0.5mg intravitreal injection. The patients would be injected at monthly intervals for the first 3 months followed by treatment on an as needed basis.
* If imatinib mesylate is safely tolerated for the first 6 weeks, the following set of 5 patients will be treated with 8 weeks of imatinib mesylate 400mg per day to be started concurrently with Lucentis 0.5mg intravitreal injection. The patients would be injected at monthly intervals for the first 3 months followed by treatment on an as needed basis.

ELIGIBILITY:
Inclusion Criteria:

* Have a BCVA letter score in the study eye between 73-24 (approximately 20/40 to 20/320) using an ETDRS chart
* Have a CNV lesion of any type in the study eye with the following characteristics as determined by fluorescein angiography:
* Evidence that CNV extends under the geometric center of the foveal avascular zone.
* The area of the CNV must occupy at least 50% of the total lesion.
* The lesion must be ≤4000 microns in greatest linear dimension (GLD)
* For occult with no classic CNV, the lesion must have presumed recent disease progression as assessed by the Investigator and defined as having at least one of the following criteria:

  * Blood associated with the lesion at baseline
  * Loss of VA in the previous 3 months defined as either
  * ≥5 letters (ETDRS equivalent) as determined by protocol refraction and protocol measurement OR- 2 or more lines using a Snellen or equivalent chart by standard examination
  * ≥10% increase in the GLD as assessed by fluorescein angiography in the previous 3 months

Exclusion Criteria:

* Have a history of prior PDT, external-beam radiation, subfoveal focal laser photocoagulation, submacular surgery, or transpupillary thermotherapy in the study eye
* Have atrophy under the center of the fovea
* Have angioid streaks, presumed ocular histoplasmosis syndrome, myopia (greater than 6 diopters), or choroidal neovascularization secondary to other causes than AMD
* Are receiving or require chronic concomitant therapy with systemic (> 5 mg) or ocular corticosteroids. Chronic concomitant therapy is defined as multiple doses taken daily for 14 or more consecutive days at any time within 6 months prior to screening
* Inability to obtain photographs, fluorescein angiography, or optical coherence tomography to document CNV, e.g. due to media opacity, allergy to fluorescein dye or lack of venous access
* Have received prior treatment with any anti-angiogenic compound or any investigational treatment (e.g. Macugen, Avastin [bevacizumab], Ruboxistaurin, Lucentis [ranibizumab], Retaane [anecortave acetate], squalamine, siRNA, VEGF-Trap etc.) for neovascular AMD
* Have the presence of fibrosis, hemorrhage, pigment epithelial detachments, tear (rip) of the retinal pigment epithelium or other hypofluorescent lesions obscuring greater than 50% of the CNV lesion
* Have any additional ocular diseases which have irreversibly compromised or follow-up could likely compromise the visual acuity of the study eye including amblyopia, anterior ischemic optic neuropathy, clinically significant diabetic macular edema, severe non-proliferative diabetic retinopathy
* Within two months prior to screening, have had intraocular surgery (including cataract surgery) in the study eye
* Within 1 month prior to screening had YAG laser in the study eye
* Have had previous intravitreal drug delivery (injection or drug device implantation) in the study eye
* Have had previous pars plana vitrectomy in the study eye
* Have systemic cancer under active treatment with chemotherapeutic agents
* Are being treated with anti-coagulants more than 325mg of aspirin per day.
* Have hepatic insufficiency as defined as an SGOT greater than the upper limit of normal or a total bilirubin 1.5 times the upper limit of normal
* Have history of congestive heart failure, myocardial infarction, transient ischemic attack and/or stroke within the last 3 months.
* Are using herbal products such as St.Johns Wort, acetaminophen (Tylenol), eruthromycin, or phenytoin (Dilatin) on a chronic basis

Min Age: 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11

PRIMARY OUTCOMES:
To determine the safety and tolerability of 0.5 mg dose of Ranibizumab in combination with a daily pill of 400mg of Imatinib Mesylate in the treatment of choroidal neovascularization secondary to age-related macular degeneration

SECONDARY OUTCOMES:
Proportion of patients losing ≤ 15 letters as measured by ETDRS visual refraction at 4 meters compared to baseline at month 3 and 6.
Proportion of patients gaining ≥ 15 letters as measured by ETDRS visual refraction at 4 meters compared to baseline at month 3 and 6
Change in central retinal thickness as measured by OCT at months 3 and 6 compared to baseline
Proportion of subjects gaining ≥ 30 letters as measured by ETDRS visual refraction at month 3 and 6
Change in leakage area seen during fluorescein angiography at 3 and 6 months as compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Spaide, M.D., Principal Investigator — Vitreous Retina Macula Consultants of New York, P.C.
Locations (1):
- Vitreous Retina Macula Consultants of New York, P.C., New York, New York, United States